CLINICAL TRIAL: NCT04405648
Title: Prevalence and Severity of Computer Vision Syndrome Among Medical Students
Brief Title: Computer Vision Syndrome Prevalence Among University Students
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Prof. Mohammed Iqbal, Assistant Professor of Ophthalmology, Sohag University
Other Study IDs: 4-8/1/2018
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Device: No

INTERVENTIONS:
Behavioral: CVS GROUP — the students will respond to CVS-F3 questionnaire to report their potential CVS complains and associated screen factors as screen-time, screen-size, screen-resolution and other factors.

SUMMARY:
CVS-F3 questionnaire will be used as an instrument to survey CVS prevalence and severity among medical students

DETAILED DESCRIPTION:
CVS-F3 is a valid questionnaire that includes 26 questions to be responded by the medical students to detect CVS complains and possible complications. The questionnaire includes questions regarding potential ocular, extra-ocular, musclo-skeletal and neuro-psychatric complains caused by CVS. Complete statistical analysis of the survey data will be done using univariate and multivariate logistic and linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* university students
* studying medicine

Exclusion Criteria:

* ocular surgery
* amblyopia
* anisometropia
* strabismus
* DM
* hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: medical students who are using screens in their medical studies or personal lives and how these screens affect their medical studies and the effect of mandated medical computer use if present on their screen-behaviour and associated risk factor
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of CVS | 1 month
  will be reorted in form of percentage (%) of students with CVS
Visual acuity | 1 month
  measurement of visual acuity using distance visual charts in logMAR measurements
Refraction | 1 month
  measurement of refractive power in diopters
Schirmer test | 1 month
  measurement of tear volume production with Schirmer test in mm unit measurements
Tear Break Up Time (TBUT) | 1 month
  measurement of tear film stability with TBUT in seconds time unit measurements
mfERG examinations | 6 months
  mfERG will be performed for the students to document the effect of CVS on retina

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Iqbal, Principal Investigator — Sohag University
Locations (2):
- Egypt (2):
  - Faculty of medicine, Sohag
  - Sohag Faculty of Medicine, Sohag

REFERENCES:
- [Derived] Iqbal M, Soliman A, Ibrahim O, Gad A. Analysis of the Outcomes of the Screen-Time Reduction in Computer Vision Syndrome: A Cohort Comparative Study. Clin Ophthalmol. 2023 Jan 7;17:123-134. doi: 10.2147/OPTH.S399044. eCollection 2023. PMID 36644605